CLINICAL TRIAL: NCT02456467
Title: HemoSonics-UVA Cardiac Surgery Clinical Study Protocol
Brief Title: HemoSonics-UVA HemoSonics-UVA Cardiac Surgery Clinical Study Protocol
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: HemoSonics LLC (Industry)
Responsible Party: Principal Investigator, Danja Groves, MD, Associate Professor, Anesthesiology, University of Virginia
Other Study IDs: 17923:
Record Dates: First submitted 2015-05-26; First posted 2015-05-28 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac Surgery Patients: Intervention: Procedure: Blood specimen collection

SUMMARY:
This study compares the results of current standard coagulation measurement devices to the Quantra System, a new device, using small amount of extra blood obtained during routine blood draws in cardiac surgery patients.

DETAILED DESCRIPTION:
HemoSonics is developing a novel POC diagnostic device, the Quantra System, to perform whole blood coagulation analysis and which is suitable for use in surgical and intensive care settings. The Quantra System employs a patented technology named sonorheometry, which was invented at the University of Virginia. Sonorheometry uses ultrasound pulses to characterize the dynamic changes in viscoelastic properties of a blood sample during coagulation and clot lysis. The initial assay performed on the Quantra System will be the surgical assay for monitoring hemostasis during major surgical procedures in adult patients.

A clinical study will be conducted to evaluate the analytical performance as well as provide a preliminary evaluation of the performance comparability of the HemoSonics' device as compared to existing coagulation monitoring technology in heart surgery. This study will be performed at HemoSonics and the University of Virginia Health System and will involve patients undergoing cardiac surgery requiring bypass.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for cardiac surgery involving bypass circuit
* Subject is older than 18 years
* Subject is willing to participate and he/she has signed a consent form

Exclusion Criteria:

* Subject is unable to provide written informed consent
* Subject is incarcerated at the time of the study
* Subject is affected by any condition that, in the opinion of the surgical team, may pose additional risks
* Patients with renal disease (defined as serum creatinine greater than 1.5 mg/dl)
* Patients with history of active liver disease
* Patients on emergency cases
* Patients on heparin anticoagulation before the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be recruited at UVA. The subject population will be representative of the local racial and ethnic population.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Clot time | 1 day
  Coagulation Function
Clot Amplitude | 1 day
  Coagulation Function

CONTACTS AND LOCATIONS:
Overall Officials: Danja Groves, MD, Principal Investigator — UVA Anesthesiology Faculty
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States